CLINICAL TRIAL: NCT04299542
Title: Percutaneous Lung Biopsy Using Cone Beam CT With Virtual Guidance: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VIR-19-11
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional Multi-detector CT (MDCT) (Active Comparator): Percutaneous lung biopsy using MDCT
  Interventions: Procedure: Percutaneous lung biopsy using conventional MDCT
- cone-beam CT (CBCT) (Active Comparator): Percutaneous lung biopsy using CBCT
  Interventions: Procedure: Percutaneous lung biopsy CBCT

INTERVENTIONS:
Procedure: Percutaneous lung biopsy using conventional MDCT — Conventional CT biopsy will be performed using a 64 slice CT scanner. A preliminary plain CT is acquired covering the entire target lesion with a skin marker, and the interventional radiologist would decide on the skin puncture site and the needle pathway. A post-procedural CT scan will be made to detect pneumothorax or pulmonary haemorrhage. All images will be archived in the picture achieving and communication system (PACS).
  Arms: conventional Multi-detector CT (MDCT)
Procedure: Percutaneous lung biopsy CBCT — CBCT guided biopsy will be performed in the angiography suite. A preliminary CBCT (DynaCT) is acquired covering the entire target lesion is first performed. Image data will be displayed and processed using Syngo iGuide system. A potential needle trajectory will be drawn from skin to lesion. Integration of the cross-sectional images and real time fluoroscopy will result in three system positions: one bull's eye view and two progression views. During fluoroscopy, the planned needle trajectory and target will be overlaid on the real time fluoroscopy image. After the needle reaches the target, another CBCT will be performed to confirm needle position. Biopsy using coaxial system and post-procedural CT scans will be performed in similar fashion as the conventional CT group.
  Arms: cone-beam CT (CBCT)

SUMMARY:
Image-guided percutaneous lung biopsy is an essential procedure in lung cancer management, where it is integral to confirming the diagnosis and determining tumour histology. An ideal percutaneous lung biopsy also needs to have a short procedure time with accurate needle placement to minimize the inherent risk of the procedure.

Since the 1970s, conventional Multi-detector CT (MDCT) has been the modality of choice in percutaneous lung biopsy. Recent research has proposed CT fluoroscopy and cone-beam CT (CBCT) as alternative methods.

Virtual guidance has been developed to improve target visibility and access for these complex cases. More specifically, it plans a potential computed 3D needle path before the procedure, using the CBCT images. This 3D path can be transposed onto real time fluoroscopic images to guide the biopsy, thus potentially improves patients' safety due to more accurate needle placement.

DETAILED DESCRIPTION:
Image-guided percutaneous lung biopsy is an essential procedure in lung cancer management, where it is integral to confirming the diagnosis and determining tumour histology. In this era of personalized medicine where knowledge of specific cellular pathways and molecular characterization relies on obtaining optimal tissue sampling, the critical question is how to obtain a high-quality biopsy tissue sample that could be processed for various pathological assessment from a single, minimally invasive percutaneous image-guided approach.

An ideal percutaneous lung biopsy also needs to have a short procedure time with accurate needle placement to minimize the inherent risk of the procedure, including the stochastic effect of radiation, and injuries to structures resulting in pneumothorax, pulmonary hemorrhage, and air embolism, which could all be potentially life threatening. Previous studies have also shown that post-biopsy haemorrhage or pneumothorax requiring chest tubes insertion had worse outcome, increased length of hospital stays, and respiratory failure.

Since the 1970s, conventional Multi-detector CT (MDCT) has been the modality of choice in percutaneous lung biopsy, which requires repeated scanning of the target lesion during the procedure and the interventional radiologist entering and leaving the CT suite after each needle adjustment. Recent research has proposed CT fluoroscopy and cone-beam CT (CBCT) as alternative methods.

Virtual guidance has been developed to improve target visibility and access for these complex cases. This involves image registration where the real-time imaging dataset is matched to a reference dataset, where the position of a device is displayed on the current imaging dataset in real time. Syngo iGuideTM is a novel navigational software which has the potential for accurate needle guidance in percutaneous biopsy. More specifically, it plans a potential computed 3D needle path before the procedure, using the CBCT images. An integrated laser crosshair is also projected onto the patient's skin to indicate the entry point and angle of the needle at no additional radiation dose to the patient and staff. This 3D path can be transposed onto real time fluoroscopic images to guide the biopsy, thus potentially improves patients' safety due to more accurate needle placement.

ELIGIBILITY:
Inclusion Criteria:

* Solitary or multiple lung lesions (solid or subsolid nodule, pulmonary infiltrate) ≥1cm

Exclusion Criteria:

* Patient <18 years old
* Patient not able to give informed consent
* Uncooperative patient who is unable to hold still or hold their breath for safe biopsy
* Lesions <1cm
* Lesions within 1cm of vital thoracic structures such as the great vessels and the mediastinum
* Peripheral lesions accessible to biopsy with ultrasound guidance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
The number of needle repositioning to reach the target | immediately after completion of procedure
  This will be recorded during procedure

SECONDARY OUTCOMES:
procedure time | immediately after completion of procedure
  This will be recorded throughout procedure
radiation dose | immediately after completion of procedure
  This will be recorded throughout procedure
complication | 1 month after completion of procedure
  observation during and after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Professor, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No